CLINICAL TRIAL: NCT05246878
Title: A Randomized, Double-Blind, Sponsor-Open, Placebo-Controlled, First In Human Study of Orally Administered EDP-235 to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses, Multiple Ascending Doses, and the Effect of Food on EDP-235 Pharmacokinetics in Healthy Participants
Brief Title: A Study of EDP-235 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EDP 235-001
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: SARS CoV 2 Infection
Keywords: First-in-Human; Single Ascending Dose; Multiple Ascending Dose; Healthy Volunteer; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — EDP-235

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- EDP-235 SAD Cohorts (Experimental): EDP-235 Dose 1, Dose 2, Dose 3, Dose 4 and Dose 5, orally, once daily in one single administration
  Interventions: Drug: EDP-235
- EDP-235 MAD Cohorts (Experimental): EDP-235 Dose 1, Dose 2 and Dose 3 orally, once daily for 7 days
  Interventions: Drug: EDP-235
- EDP-235 SAD Placebo Cohorts (Placebo Comparator): Matching placebo, orally, once daily in one single administration
  Interventions: Drug: Placebo
- EDP-235 MAD Placebo Cohorts (Placebo Comparator): Matching placebo, orally, once daily for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EDP-235 — Oral administration
  Arms: EDP-235 MAD Cohorts; EDP-235 SAD Cohorts
Drug: Placebo — Placebo to match EDP-235, oral administration
  Arms: EDP-235 MAD Placebo Cohorts; EDP-235 SAD Placebo Cohorts

SUMMARY:
This study is a randomized, double-blind, placebo-controlled study. It will assess the safety, tolerability, and pharmacokinetics of orally administered single and multiple doses of EDP-235 in healthy adult subjects.

DETAILED DESCRIPTION:
The first phase assesses single ascending doses of EDP-235 or placebo in healthy subjects. A "fasted" and "fed" two-part cohort will also assess food effect.

The second phase assesses multiple ascending doses of EDP-235 or placebo for 7-days in healthy subjects.

Each cohort within each phase will enroll a total of 8 subjects who will be randomized to receive EDP-235 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document signed and dated by the subject.
* Healthy male and female subjects of any ethnic origin between the ages of 18 and 65 years, inclusive.

Exclusion Criteria:

* Clinically relevant evidence or history of illness or disease.
* Infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) at screening and infection with SARS-CoV-2 at the Day -1 visit
* Pregnant or nursing females.
* History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection.
* A positive urine drug screen at screening or Day -1.
* Current tobacco smokers or use of tobacco within 3 months prior to screening.
* Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy).
* History of regular alcohol consumption.
* Receipt of any vaccine, an investigational agent or biological product within 28 days or 5 times the t½, whichever one is longer, prior to first dose.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Safety measured by adverse events | Up to 8 Days in HV SAD Cohorts
Safety measured by adverse events | Up to 14 Days in HV MAD Cohorts

SECONDARY OUTCOMES:
Cmax of EDP-235 | Up to 5 Days in HV SAD Cohorts
AUC of EDP-235 | Up to 5 Days in HV SAD Cohorts
Cmax of EDP-235 | Up to 11 Days in HV MAD Cohorts
AUC of EDP-235 | Up to 11 Days in HV MAD Cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (1):
- Pharmaceutical Research Associates, Inc.,, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No